CLINICAL TRIAL: NCT01085669
Title: Infection Rate of VEPTR-Implants in Children With Severe Spinal and Thoracic Deformities
Brief Title: Infection Rate of Vertical Expandable Prosthetic Titanium Rib Implants (VEPTR)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: University Children's Hospital Basel (Other)
Responsible Party: PD Dr. Carol-C. Hasler, Head Spine Surgery, Orthopaedic Department, University Children´s Hospital Basel
Other Study IDs: EKBB 304/09
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2010-03-12 (Estimated); Status verified 2010-03

CONDITIONS: Infection
Keywords: Infection rate of VEPTR-Implants; VEPTR. Vertical Expandable; Prosthetic Titanium Rib
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VEPTR patients: Children treated with VEPTR Implants for severe spinal or thoracic deformities
  Interventions: Device: Microbiological analysis of retained VEPTR Implants

INTERVENTIONS:
Device: Microbiological analysis of retained VEPTR Implants — Implants have to be adapted every half a year, the retained implants during revision are analysed for biological colonization.

SUMMARY:
The study is conducted to analyse the infection rate in children treated with VEPTR-Implants for severe spine or thoracic deformities.

DETAILED DESCRIPTION:
Spinal and thoracic deformities in children can be treated with vertical expandable prosthetic titanium ribs (VEPTR©, Synthes GmbH®) to stimulate thoracic and spinal growth. With these implants children's symptoms and conditions can be slowed, halted or even reversed. Because of the dynamic character of the deformity and the growth of the children, the implants have to be lengthened about every half a year. With each operation there is a small risk of infection, which might increase with number of previous surgeries. Implant associated infections are often not clinical apparent and only found in microbiological analysis. To objectify the infection rate, identify potential precursors of infections and the relevance of asymptomatic infections in children with these implants a prospective study is conducted.

ELIGIBILITY:
Inclusion Criteria:

* all patients admitted at the University Children's Hospital Basel in whom a VEPTR©-implant or parts of it will be removed.

Exclusion Criteria:

* obvious contamination of an explanted component occurred in the operating room.

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with severe spinal or throacic deformities treates with VEPTR-implants. In these patients the implant has to be revised every half a year due to grow and achieved correction.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-12 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Infection rate of VEPTR Implants | two years

CONTACTS AND LOCATIONS:
Locations (1):
- Orthopaedic Department, University Children´s Hospital Basel, Basel, Switzerland